CLINICAL TRIAL: NCT05026762
Title: The Impact of Social Phone Calls With Isolated Older Adults Receiving Protective Services for Abuse, Neglect and/or Exploitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: UTHealth Consortium on Aging (Unknown)
Responsible Party: Principal Investigator, Gabrielle Marie Hoyumpa, Student, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-21-0411
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Senior Abuse
Keywords: depression; anxiety; loneliness; isolation; adult protective services
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — Following the collection of the baseline data, the study participant will be assigned to a volunteer(medical student) to begin the social phone calls. The first phone call will be scheduled to occur within one week of the consent and baseline assessments. A minimum of one social phone call will occur each week for 6-weeks. Each phone call is expected to last up to 1 hour.The calls will be unstructured and designed simply to engage in conversation with the participant. The length of the phone calls, days and times will be recorded by the volunteer along with a short journal entry describing the conversation topics and any information that stood out to the volunteer.At the end of the 6-weeks phone calls, a group session will be held with the volunteers to engage in a debriefing and narrative medicine session.

SUMMARY:
The purpose of this study is to see the the impact of social visits, through weekly phones calls, on quality of life outcomes of depression, anxiety, loneliness, isolation and self-rated health for older adults visited by Adult Protective Services (APS) for abuse, neglect and/or exploitation (ANE) and to also to determine the benefit of these conversations on the medical student's perspective of aging and ANE.

ELIGIBILITY:
Inclusion Criteria:

* recently visited by Texas Adult Protective Services for Abuse, Neglect and/or Exploitation
* living in Harris County or a surrounding county serviced by APS District 6
* substantiated elder mistreatment (i.e. psychological abuse, financial exploitation, sexual abuse, neglect, physical abuse) and/or self neglect
* provide a signed or verbal release agreeing to be contacted by the volunteers
* able to provide verbal consent to participate in the study

Exclusion Criteria:

* significant cognitive impairment or incapacity as determined by their inability to complete the consent steps
* Non-English-speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Social isolation as assessed by the patient-reported outcomes measurement information system (PROMIS) Social Isolation Scale | Baseline, 6 week follow up
  This is a 4 item questionnaire and each question is scored from 1(never) to 5(always) a higher number indicating more isolation
Change in Anxiety as assessed by the Geriatric Anxiety Scale | Baseline, 6 week follow up
  This is a 10 item questionnaire and each question is scored form 0(not at all) to 3(most of the time),a higher number indicating more anxiety
Change in Depression as assessed by the Geriatric Depression Scale Short Form | Baseline, 6 week follow up
  This is a 15 item questionnaire and each is answered either yes or no. One point is given for No to question 1, 5, 7, 11, 13 and one point for Yes to other questions.
  Normal ± 2 Mildly Depressed 7 ± 3 Very Depressed 12 ± 2
Change in Loneliness as assessed by the University of California Los Angeles (UCLA ) Loneliness Scale | Baseline, 6 week follow up
  A 20-item scale that measures the subjective experience of loneliness on a four-point Likert scale. Participants rate each item as either O (I often feel this way),S (I sometimes feel this way), R (I rarely feel this way), N (I never feel this way).
Change in perceived general health as assessed by the Self-Rated Health Question | Baseline, 6 week follow up
  The participant will rate their health as excellent, very good, good, fair or poor

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle M Hoyumpa, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No